CLINICAL TRIAL: NCT04176731
Title: Prepivotal Evaluation of the Safety and Effectiveness of the Omnipod Horizon™ Automated Glucose Control System in Patients With Type 1 Diabetes
Brief Title: Prepivotal Omnipod Horizon™ Automated Glucose Control System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insulet Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Horizon™ Prepivotal Study
Record Dates: First submitted 2019-11-15; First posted 2019-11-25 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: T1D; Omnipod
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: This is a single-arm, multi-center, prospective clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): All subjects wearing the Omnipod Horizon™ Automated Glucose Control System using the closed-loop algorithm
  Interventions: Device: Omnipod Horizon™ Automated Glucose Control System

INTERVENTIONS:
Device: Omnipod Horizon™ Automated Glucose Control System — The Omnipod Horizon™ Automated Glucose Control System will provide automated insulin delivery

SUMMARY:
Subjects will undergo a 14-day outpatient, standard therapy phase during which sensor and insulin data will be collected. This will be followed by a 14-day hybrid closed-loop phase conducted in both a hotel/rental house setting and outpatient setting.

DETAILED DESCRIPTION:
The study schedule will consist of a standard therapy data collection phase followed by a hybrid closed-loop phase.

Subjects will undergo a 14-day outpatient, standard therapy phase during which sensor and insulin data will be collected. Subjects, or their caregivers, will manage their diabetes at home per their usual routine using the study continuous glucose monitoring system (CGM) and remain on current multiple daily injections (MDI) or pump therapy. This will be followed by a 14-day hybrid closed-loop phase conducted in both a hotel/rental house setting and an outpatient setting.

The hybrid closed-loop phase will begin on Study Day 1.

During the hybrid closed-loop phase, subjects will be divided into two groups. The first group of subjects will commence the hybrid closed-loop phase in the hotel/rental house setting. On Study Day 3, subjects will transition to an outpatient setting for the remaining 12 days. After all subjects from the first group have completed the 2-day hotel/rental house phase, the second group of subjects may commence the hybrid closed-loop phase in an outpatient setting for 14-days.

During the hybrid closed-loop phase, all subjects will participate in specific target blood glucose (BG) challenges.

After each subject in the prepivotal study has successfully completed 14-days of hybrid-closed-loop, they may immediately transition to and enroll in the pivotal study.

ELIGIBILITY:
Inclusion Criteria:

1. Age at time of consent/assent 6-70 years
2. Subjects aged < 18 years must be living with parent/legal guardian
3. Diagnosed with type 1 diabetes for at least 6 months. Diagnosis is based on investigator's clinical judgment.
4. Deemed appropriate for pump therapy per investigator's assessment taking into account previous history of severe hypoglycemic and hyperglycemic events, and other comorbidities
5. Investigator has confidence that the subject can successfully operate all study devices and is capable of adhering to the protocol
6. Willing to use only the following types of insulin during the study: Humalog, Novolog, Admelog, or Apidra during the study
7. Must be willing to set target glucose between 130-150 mg/dL each for approximately 72-hours on predefined days during the hybrid closed-loop phase
8. Must be willing to extend their participation into the pivotal study if they continue to meet the protocol criteria
9. Willing to wear the system continuously throughout the study
10. A1C <10% at screening visit
11. Must be willing to use the Dexcom App on the Omnipod Horizon™ PDM as the sole source of Dexcom data (with the exception of the Dexcom Follow App) during the hybrid closed-loop phase
12. Subjects scoring ≥ 4 on the Clarke Questionnaire must agree to have an overnight companion, defined as someone who resides in the same home or building as the study subject and who can be available overnight
13. Able to read and speak English fluently
14. Subject must be in an AT&T covered area
15. Willing and able to sign the Informed Consent Form (ICF) and/or has a parent/guardian willing and able to sign the ICF. Assent will be obtained from pediatric and adolescent subjects aged < 18 years per State requirements.

Exclusion Criteria:

1. A medical condition, which in the opinion of the investigator, would put the subject at an unacceptable safety risk
2. History of severe hypoglycemia (as defined in Section 11.3.3) in the past 6 months
3. History of DKA (as defined in Section 11.3.4) in the past 6 months, unrelated to an intercurrent illness, infusion set failure or initial diagnosis
4. Diagnosed with sickle cell disease
5. Diagnosed with hemophilia or any other bleeding disorders
6. Plans to receive blood transfusion over the course of the study
7. Currently diagnosed with anorexia nervosa or bulimia
8. Acute or chronic kidney disease (e.g. estimated GFR < 45) or currently on hemodialysis
9. History of adrenal insufficiency
10. Has taken oral or injectable steroids within the past 8 weeks or plans to take oral or injectable steroids during the course of the study
11. Unable to tolerate adhesive tape or has any unresolved skin condition in the area of sensor or pump placement
12. Plans to use insulin other than U-100 insulin intended for use in the study device during the course of the study
13. Use of non-insulin anti-diabetic medication other than metformin (e.g. GLP1 agonist, SGLT2 inhibitor, DPP-4 inhibitor, pramlintide)
14. Current or known history of coronary artery disease that is not stable with medical management, including unstable angina, or angina that prevents moderate exercise despite medical management, or a history of myocardial infarction, percutaneous coronary intervention, or coronary artery bypass grafting within the previous 12 months.
15. For subjects >50 years old or with diabetes duration >20 years, abnormal electrocardiogram consistent with increased risk of arrhythmia, ischemia, or prolonged QTc interval (> 450 ms)
16. Thyroid Stimulating Hormone (TSH) is outside of normal range with clinical signs of hypothyroidism or hyperthyroidism
17. Pregnant or lactating, or is a woman of childbearing potential and not on acceptable form of birth control (acceptable includes abstinence, condoms, oral/injectable contraceptives, IUD or implant)
18. Participation in another clinical study using an investigational drug or device within the preceding 30-days or intends to participate during the study period
19. Unable to follow clinical protocol for the duration of the study or is otherwise deemed unacceptable to participate in the study per the investigator's clinical judgment.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Buckingham, MD, Study Chair — Stanford University; Sue Brown, MD, Study Chair — University of Virginia
Locations (6):
- United States (6):
  - Stanford University, Palo Alto, California
  - University of Colorado Denver, Denver, Colorado
  - Atlanta Diabetes, Atlanta, Georgia
  - International Diabetes Center, Saint Louis Park, Minnesota
  - Mount Sinai, New York, New York
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.8 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.6 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Severe Hypoglycemia
Description: Measure of serious device-related adverse events
Time Frame: hybrid closed-loop (14 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 36
Participants | 0

2. Primary Outcome: Proportion of Subjects With Diabetic Ketoacidosis (DKA)
Description: Measure of serious device-related adverse events
Time Frame: hybrid closed-loop (14 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 36
Participants | 0

3. Primary Outcome: Percentage of Time in Range 70-180 mg/dL During Target Blood Glucose Challenge Days of Hybrid Closed Loop Phase (Days 1-9) and Standard Therapy Period (14 Days)
Description: Percentage of time in range 70-180 mg/dL
Time Frame: hybrid closed-loop (9 days) compared to standard therapy (14 days)
Measure: Mean (Standard Deviation); unit: Overall Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 36
Overall Percent Time in Range
  Day Time ST | 58 (17.1)
  Day Time HCL | 62.2 (9.6)
  Night Time ST | 59.2 (16.4)
  Night Time HCL | 71.2 (14.0)
  Overall ST | 58.3 (16.2)
  Overall HCL | 64.4 (8.2)

4. Primary Outcome: Percentage of Time in Range 70-180 mg/dL During Non-Challenge Days of Hybrid Closed Loop Phase (Days 10-14) and Standard Therapy Period (14 Days)
Description: Percentage of time in range 70-180 mg/dL
Time Frame: hybrid closed-loop (5 days) compared to standard therapy (14 days)
Measure: Mean (Standard Deviation); unit: Overall Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 36
Overall Percent Time in Range
  Day Time ST | 58.0 (17.1)
  Day Time HCL | 67.2 (11.9)
  Night Time ST | 59.2 (16.4)
  Night Time HCL | 72.8 (18.2)
  Overall ST | 58.3 (16.2)
  Overall HCL | 68.7 (11.3)

5. Primary Outcome: Percentage of Time in Range 70-180 mg/dL During Overall (Days 1-14) and Standard Therapy Period (14 Days)
Description: Percentage of time in range 70-180 mg/dL
Time Frame: hybrid closed-loop (14 days) compared to standard therapy (14 days)
Measure: Mean (Standard Deviation); unit: Overall Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 36
Overall Percent Time in Range
  Day Time ST | 58.0 (17.1)
  Day Time HCL | 63.9 (8.3)
  Night Time ST | 59.2 (16.4)
  Night Time HCL | 71.1 (13.3)
  Overall ST | 58.3 (16.2)
  Overall HCL | 65.8 (7.3)

6. Secondary Outcome: Mean Glucose
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: hybrid closed-loop (14 days) compared to the standard therapy (14 days) during the day, overnight, and overall
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment
Number analyzed (Participants) | 36
mg/dL
  Day Time ST | 172.8 (29.8)
  Day Time HCL | 168.4 (12.7)
  Night Time ST | 165.8 (28.4)
  Night Time HCL | 163.0 (16.2)
  Overall ST | 171.2 (27.7)
  Overall HCL | 167.0 (11.5)

7. Secondary Outcome: Time in Range 70-180 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: hybrid closed-loop (14 days) compared to the standard therapy (14 days) during the day, overnight, and overall
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 36
Percent Time in Range
  Day Time ST | 58.0 (17.1)
  Day Time HCL | 63.9 (8.3)
  Night Time ST | 59.2 (16.4)
  Night Time HCL | 71.1 (13.3)
  Overall ST | 58.3 (16.2)
  Overall HCL | 65.8 (7.3)

8. Secondary Outcome: Time in Range 70-140 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: hybrid closed-loop (14 days) compared to the standard therapy (14 days) during the day, overnight, and overall
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 36
Percent Time in Range
  Day Time ST | 35.7 (15.6)
  Day Time HCL | 33.2 (6.7)
  Night Time ST | 37.8 (16.7)
  Night Time HCL | 35.3 (12.8)
  Overall ST | 36.2 (15.2)
  Overall HCL | 33.8 (6.9)

9. Secondary Outcome: Percentage of Time >180 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: hybrid closed-loop (14 days) compared to the standard therapy (14 days) during the day, overnight, and overall
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 36
Percent Time in Range
  Day Time ST | 39.5 (18.4)
  Day Time HCL | 35.1 (8.5)
  Night Time ST | 36.6 (17.7)
  Night Time HCL | 27.8 (13.4)
  Overall ST | 38.8 (17.2)
  Overall HCL | 33.3 (7.6)

10. Secondary Outcome: Percentage of Time ≥250 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: hybrid closed-loop (14 days) compared to the standard therapy (14 days) during the day, overnight, and overall
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 36
Percent Time in Range
  Day Time ST | 14.6 (10.7)
  Day Time HCL | 9.1 (6.1)
  Night Time ST | 12.6 (10.5)
  Night Time HCL | 6.5 (6.6)
  Overall ST | 14.1 (9.9)
  Overall HCL | 8.5 (5.4)

11. Secondary Outcome: Percentage of Time ≥300 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: hybrid closed-loop (14 days) compared to the standard therapy (14 days) during the day, overnight, and overall
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 36
Percent Time in Range
  Day Time ST | 5.6 (5.9)
  Day Time HCL | 2.4 (2.4)
  Night Time ST | 4.6 (5.8)
  Night Time HCL | 2.0 (3.2)
  Overall ST | 5.4 (5.3)
  Overall HCL | 2.3 (2.2)

12. Secondary Outcome: Percentage of Time <70 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: hybrid closed-loop (14 days) compared to the standard therapy (14 days) during the day, overnight, and overall
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 36
Percent Time in Range
  Day Time ST | 2.4 (2.6)
  Day Time HCL | 1.0 (1.1)
  Night Time ST | 4.2 (5.2)
  Night Time HCL | 0.5 (1.3)
  Overall ST | 2.9 (3.0)
  Overall HCL | 0.9 (1.1)

13. Secondary Outcome: Percentage of Time <54 mg/dL
Description: Glucose metric from study continuous glucose monitoring system (CGM)
Time Frame: hybrid closed-loop (14 days) compared to the standard therapy (14 days) during the day, overnight, and overall
Measure: Mean (Standard Deviation); unit: Percent Time in Range
Arm/Group | Treatment
Number analyzed (Participants) | 36
Percent Time in Range
  Day Time ST | 0.5 (0.7)
  Day Time HCL | 0.1 (0.3)
  Night Time ST | 1.1 (1.8)
  Night Time HCL | 0.1 (0.4)
  Overall ST | 0.6 (0.9)
  Overall HCL | 0.1 (0.3)

14. Secondary Outcome: Standard Deviation of Glucose (mg/dL)
Description: Glucose metric from study continuous glucose monitoring system (CGM)-measured glucose variability with the standard deviation (SD)
Time Frame: hybrid closed-loop (14 days) compared to the standard therapy (14 days) during the day, overnight, and overall
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment
Number analyzed (Participants) | 36
mg/dL
  Day Time ST | 62.9 (14.7)
  Day Time HCL | 53.4 (9.5)
  Night Time ST | 60.5 (17.8)
  Night Time HCL | 45.0 (14.2)
  Overall ST | 63.3 (14.9)
  Overall HCL | 52.3 (9.4)

15. Secondary Outcome: Coefficient of Variation
Description: Glucose metric from study continuous glucose monitoring system (CGM)-measured glucose variability with the coefficient of variation (CV)
Time Frame: hybrid closed-loop (14 days) compared to the standard therapy (14 days) during the day, overnight, and overall
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Treatment
Number analyzed (Participants) | 36
Percent
  Day Time ST | 36.3 (5.0)
  Day Time HCL | 31.6 (4.4)
  Night Time ST | 36.5 (9.2)
  Night Time HCL | 27.3 (7.2)
  Overall ST | 36.9 (5.9)
  Overall HCL | 31.2 (4.6)

16. Secondary Outcome: Glucose Management Indicator (GMI) Based on Overall Mean Glucose
Description: Measurement of glucose management using overall glucose averages
Time Frame: hybrid closed-loop (14 days) compared to the standard therapy (14 days)
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Treatment
Number analyzed (Participants) | 36
Percent
  Day Time ST | 7.4 (0.7)
  Day Time HCL | 7.3 (0.3)
  Night Time ST | 7.3 (0.7)
  Night Time HCL | 7.2 (0.4)
  Overall ST | 7.4 (0.7)
  Overall HCL | 7.3 (0.3)

17. Secondary Outcome: Percentage of Time in Hybrid Closed-loop as Proportion of Overall Device Usage Time
Description: Measure of system usage
Time Frame: hybrid closed-loop (14 days)
Measure: Mean (Standard Deviation); unit: Percent Time Spent
Arm/Group | Treatment
Number analyzed (Participants) | 36
Percent Time Spent
  Automated Mode | 97.3 (3)
  Manual Mode | 2.1 (2.2)

18. Secondary Outcome: Total Daily Insulin (TDI) (Units, Units/kg)
Description: Measure of insulin requirements
Time Frame: hybrid closed-loop (14 days) compared to the standard therapy (14 days)
Measure: Mean (Standard Deviation); unit: units/kg
Arm/Group | Treatment
Number analyzed (Participants) | 36
units/kg
  ST | 39.5 (13.5)
  HCL | 37.0 (14.5)

19. Secondary Outcome: Total Daily Basal Insulin (Units, Units/kg)
Description: Measure of insulin requirements
Time Frame: hybrid closed-loop (14 days) compared to the standard therapy (14 days)
Measure: Mean (Standard Deviation); unit: units/kg
Arm/Group | Treatment
Number analyzed (Participants) | 36
units/kg
  ST | 20.7 (10.3)
  HCL | 17.5 (7.6)

20. Secondary Outcome: Total Daily Bolus Insulin (Units, Units/kg)
Description: Measure of insulin requirements
Time Frame: hybrid closed-loop (14 days) compared to the standard therapy (14 days)
Measure: Mean (Standard Deviation); unit: units/kg
Arm/Group | Treatment
Number analyzed (Participants) | 36
units/kg
  ST | 19.4 (8.5)
  HCL | 19.5 (7.8)

ADVERSE EVENTS:
Time Frame: First day of standard therapy to the last day in hybrid closed loop phase, average of 28 days.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 4/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=36)
Skin Infection (Skin and subcutaneous tissue disorders) | 1
Ketosis (Metabolism and nutrition disorders) | 1
Prolonged Hyperglycemia (Endocrine disorders) | 1
Shoulder problem (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT04176731/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/31/NCT04176731/SAP_001.pdf